CLINICAL TRIAL: NCT07226830
Title: Quantification of Change in MG Disease Activity in Individuals With Generalized Myasthenia Gravis (gMG) After Administration of VYVGART® or VYVGART Hytrulo® Using BioDigit MG
Acronym: BioDigit MG-03
Status: Not yet recruiting | Type: Observational
Sponsor: BioSensics (Industry)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BioDigit MG-03
Record Dates: First submitted 2025-11-07; First posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Myasthenia Gravis Generalized
Keywords: myasthenia gravis; digital health; wearable sensors
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- gMG group: All participants meeting the study inclusion criteria will be assigned to this group to complete the study activities

SUMMARY:
Evaluate the feasibility of using digital health technologies to monitor disease symptoms over time in individuals with gMG who are initiating treatment with VYVGART® or VYVGART Hytrulo®.

Study subjects will be screened and enrolled at Massachusetts General Brigham Hospital to participate in this 16 week observational study.

Study subjects will be asked to wear multiple wearable sensors to monitor their physical activity and PPG during daily activities. Participants will also complete speech, video, and ePRO and eCOA digital assessments at home and during study visits.

The primary objective of this observational clinical study is to remotely evaluate MG-specific outcomes using digital health technologies in individuals with gMG during two treatment cycles with VYVGART® or VYVGART Hytrulo®.

DETAILED DESCRIPTION:
MG is a chronic autoimmune neuromuscular disease characterized by fluctuating muscle weakness that interferes with activities of daily living. Ocular, facial, swallowing, neck, limb and breathing muscles can be affected. The prevalence of MG is estimated at approximately 60,000 patients in the United States. MG symptoms are currently assessed in person through a careful history and physical exam by a neuromuscular disease expert. This is time-consuming, costly, and poses challenges in a chronic disease with fluctuating symptoms, where patients may not demonstrate any abnormality at the time of in-clinic assessment. The principal means of measuring disease severity are specific scales such as the MGC, QMG and the MG Manual Muscle Testing (MMT) scales. Although valuable, these scales are subjective and require training to administer correctly. Additionally, they provide only snapshot of a patient's disease and do not adequately reflect the spectrum of fluctuating weakness, which is a hallmark of MG. Wearable sensors and digital health technologies could enable objective, sensitive, continuous assessment of physical activity as well as motor and ocular impairments in individuals with MG.

BioSensics LLC (Newton, MA) is a medical device company specializing in wearable sensors and digital health technology for healthcare. BioSensics LLC offers a wearable sensor system and digital health solution for long-term remote monitoring of motor performance during everyday life.

This is an analytic observational study following participants over the course of 16 weeks. Subjects diagnosed with gMG who are initiating treatment with VYVGART® or VYVGART Hytrulo® will be screened and recruited to participate in this non--interventional study.

In addition to standard clinical assessments, the study will leverage BioDigit MG to remotely collect high-frequency wearable and digital health data from participants in their home environments during two treatment cycles with VYVGART® or VYVGART Hytrulo®. The frequency of at-home data collection is increased during the first 2 weeks and last 2 weeks of each treatment cycle to provide a more granular data both the initial phase (first two weeks) and the last two weeks of each treatment cycle. A key objective of the project is to measure changes in disease symptoms using both patient reported outcomes (PROs) and digital measures in individuals with gMG during the treatment cycles. The investigators will also evaluate if the combination of sensors-derived and digital measures from the BioDigit MG serves as a significant early predictor of the standard clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of autoimmune MG with or without history of thymoma
* MGFA severity class IIa/b, IIIa/b or IVa/b at the screening visit
* Diagnosed gMG through one or more of the following:
* Positive acetylcholine receptor antibody (AChR Ab) test, or
* Abnormal neuromuscular transmission demonstrated by single-fiber electromyography (SFEMG) or repetitive nerve stimulation (RNS), or
* Documented positive response to standard MG therapies (e.g., AChE inhibitors, IVIG/PLEX, FcRn antagonists or C5 inhibitors)
* Currently initiating treatment with VYVGART® or VYVGART Hytrulo®
* Physically and cognitively able to provide informed consent and adhere to the study procedures, as determined by the investigator.
* Ambulatory, defined as the ability to walk at least 10 meters independently, with or without the use of an assistive device.
* Speaks and reads English fluently

Exclusion Criteria:

* Inability to perform essential activities of daily living required for independent living, such as dressing, bathing, toileting, or eating without assistance.
* Presence of neurological or orthopedic conditions unrelated to MG that, in the investigator's judgment, significantly impair gait or daily functioning.
* Any clinically significant medical, laboratory, or psychiatric condition that, in the opinion of the investigator, could interfere with study participation or data integrity.
* Current residence in a long-term care or institutional facility (e.g., nursing home, skilled nursing facility), receipt of hospice care, or incarceration.
* MGFA severity classification of Class I or Class V (myasthenic crisis). Pregnant or breastfeeding women.
* Concurrent participation in another interventional clinical trial (participation in observational studies, biomarker studies, or registries is permitted).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with gMG with MGFA severity class IIa/b, IIIa/b or IVa/b who are initiating treatment with VYVGART® or VYVGART Hytrulo®
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in total score of Myasthenia Gravis Activities of Daily Living (MG-ADL) Questionnaire from baseline to 16 weeks | From baseline to 16 weeks.
  Scores for the MG-ADL range from 0-24. A lower score represents a better outcome and a higher score is a worse outcome. Collected 11 times at home, and once at each clinical visit.
Change in total score of Myasthenia Gravis Quality of Life - Revised (MGQoL-15r) from baseline to 16 weeks | From baseline to 16 weeks.
  Scores for the MGQoL-15R range from 0-30. A lower score represents a better outcome and a higher score is a worse outcome. Collected 11 times at home, and once at each clinical visit.
Change in total score of Quality of Life in Neurological Disorders - Fatigue (Neuro-QoL Fatigue) from baseline to 16 weeks | From baseline to 16 weeks. Collected 11 times at home, and once at each clinical visit.
  Scores for the Neuro-QoL Fatigue range from 8-40. A lower score represents a better outcome and a higher score is a worse outcome.
Change in daily walking duration during activities of daily living from baseline to 16 weeks as measured by the PAMSys pendant | From baseline to 16 weeks.
  Daily walking duration (hours) will be measured by the PAMSys pendant. PAMSys is a FDA-listed Class II wearable device for measuring physical activity and posture during activities of daily living. PAMSys will be worn for 1 week before the baseline, Visit 2 (approximately week 8) , and Visit 3 (approximately week 16)
Change in daily number of sit to stand transitions (count) during activities of daily living from baseline to 16 weeks as measured by the PAMSys pendant | From baseline to week 16.
  Daily number of sit to stand transitions will be measured by the PAMSys pendant. PAMSys is a FDA-listed Class II wearable device for measuring physical activity and posture during activities of daily living. PAMSys will be worn for 1 week before the baseline, Visit 2 (approximately week 8), and Visit 3 (approximately week 16).

SECONDARY OUTCOMES:
Change in intelligibility when reading a standard Rainbow passage from baseline to 16 weeks as measured by BioDigit Speech | From baseline to 16 weeks.
  Speech data will be collected from participants while reading a standard Rainbow passage. Speech data will be collected 11 times using the at-home platform. Speech data will also be collected at each clinical visit.
  BioDigit Speech, an automatic speech analysis software, will be used to analyze the collected speech data to calculate intelligibility of speech during reading a standard Rainbow passage.
Change in Marginal Reflex Distance-1 during the upward gaze test as measured by BioDigit Video from baseline to 16 weeks | From baseline to 16 weeks.
  Video data will be collected from participants while performing a standard upward gaze test. Video data will be collected 11 times using the at-home platform. Video data will also be collected at each clinical visit.
  BioDigit Video, an automatic video analysis software, will be used to analyze the collected video data to calculate Marginal Reflex Distance-1 during the upward gaze test.
Change in total score of the Myasthenia Garvis Composite (MGC) questionnaire from baseline to 16 weeks | From baseline to 16 weeks.
  Scores for the MGC range from 0-50. A lower score represents a better outcome and a higher score is a worse outcome. Collected once at each clinical visit.
Change in total score of the Quantitative Myasthenia Gravis (QMG) scale from baseline to 16 weeks | From baseline to 16 weeks.
  Scores for the QMG range from 0-39. A lower score represents a better outcome and a higher score is a worse outcome. Collected once at each clinical visit.

OTHER OUTCOMES:
Change in daily mean heart rate (beats per minute or BPM) during activities of daily living from baseline to 16 weeks as measured by the Samsung Galaxy watch | From baseline to 16 weeks.
  Heart rate will be measured during activities of daily living using the Samsung Galaxy watch. Samsung Galaxy watch will be worn continuously from 1 week prior to baseline until the end of study visit.
Change in forced vital capacity during a standard spirometer breathing test from baseline to 16 weeks as measured by a FDA-listed spirometer | From baseline to 16 weeks.
  Forced vital capacity (FVC) will be measured directly by the spirometer during a standard breathing assessment. The FVC will be measured in Litres. FVC will be collected 11 times at home, and once at each clinical visit.
Change in mean articulatory rate when reading a standard Rainbow passage from baseline to 16 weeks as measured by BioDigit Speech | From baseline to 16 weeks.
  Speech data will be collected from participants while reading a standard Rainbow passage. Speech data will be collected 11 times using the at-home platform. Speech data will also be collected at each clinical visit.
  BioDigit Speech, an automatic speech analysis software, will be used to analyze the collected speech data to calculate intelligibility of speech during reading a standard Rainbow passage.
Change in mean eye aspect ratio during the upward gaze test as measured by BioDigit Video from baseline to 16 weeks | Baseline to 16 weeks.
  Video data will be collected from participants while performing a standard upward gaze test. Video data will be collected 11 times using the at-home platform. Video data will also be collected at each clinical visit.
  BioDigit Video, an automatic video analysis software, will be used to analyze the collected video data to calculate eye aspect ratio during the upward gaze test.
Change in daily mean heart rate variability during activities of daily living from baseline to 16 weeks as measured by the Samsung Galaxy watch | From baseline to 16 weeks.
  Heart rate variability will be measured during activities of daily living using the Samsung Galaxy watch. Samsung Galaxy watch will be worn continuously from 1 week prior to baseline until the end of study visit

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Neuromuscular Diagnostic Center, Boston, Massachusetts, United States